CLINICAL TRIAL: NCT04885283
Title: Factors Affecting the Time to Start Postoperative Chemotherapy in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, Assoc Prof, Inonu University
Other Study IDs: 2021/368
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: the Time to Start Postoperative Chemotherapy
Keywords: Laparoscopy; overall survival; local recurrence; tumor; chemotherapy; colorectal cancer
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancers are common tumors and have undergone a great change in the last 20 years in terms of treatment principles. Significantly improved results in local recurrence and overall survival have begun to be obtained with chemotherapy protocols given after surgery, which is the main element of the treatment system (1). It is known that postoperative chemotherapy protocols are commonly given within 6-8 weeks and this period is optimal. However, it was found that this period was prolonged in approximately 20% of these patients in the methanalysis performed (2). It has been shown that delay in applied chemotherapy causes a decrease in overall survival (3,4). The factors causing this delay have not been adequately examined in the literature. It is necessary to investigate these factors that affect the overall survival outcomes, which are the main pillars of treatment principles, and to regulate the factors that have the opportunity to improve.

In this study, our aim is to investigate the perioperative (preop-perop-postop) factors affecting the duration of postoperative chemotherapy initiation in patients with colorectal cancer treated in our hospital.

ELIGIBILITY:
Inclusion Criteria:

patients who underwent colorectal resection

Exclusion Criteria:

patients with missing data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent colorectal resection at General Surgery Clinic in Kayseri state hospital between January 2013 and July 2020
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Time to Start Postoperative Chemotherapy | 3 months
  time elapsed to start chemotherapy after the operation

CONTACTS AND LOCATIONS:
Overall Officials: ersin Gundogan, Assoc Prof, Study Director — Health Science University- Kayseri State Hospital
Locations (1):
- Health science University - Kayseri State Hospital, Kocasinan, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No